CLINICAL TRIAL: NCT04549259
Title: Testing a Multi-Component Intervention to Improve Health Outcomes and Quality of Life Among Rural Older Adults Living With HIV
Brief Title: Multi-Component Intervention to Improve Health Outcomes and Quality of Life Among Rural Older Adults Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jennifer Walsh, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R56NR019443 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Social Support + Stigma Reduction + SBCM + Tech Detailing (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: HIV Stigma Reduction; Behavioral: Strengths-Based Case Management (SBCM); Behavioral: Personalized Technology Detailing
- Social Support + Stigma Reduction + SBCM (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: HIV Stigma Reduction; Behavioral: Strengths-Based Case Management (SBCM)
- Social Support + Stigma Reduction + Technology Detailing (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: HIV Stigma Reduction; Behavioral: Personalized Technology Detailing
- Social Support + Stigma Reduction (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: HIV Stigma Reduction
- Social Support + SBCM + Technology Detailing (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: Strengths-Based Case Management (SBCM); Behavioral: Personalized Technology Detailing
- Social Support + SBCM (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: Strengths-Based Case Management (SBCM)
- Social Support + Technology Detailing (Experimental)
  Interventions: Behavioral: Group-Based Social Support; Behavioral: Personalized Technology Detailing
- Social Support (Experimental)
  Interventions: Behavioral: Group-Based Social Support
- Stigma Reduction + SBCM + Technology Detailing (Experimental)
  Interventions: Behavioral: HIV Stigma Reduction; Behavioral: Strengths-Based Case Management (SBCM); Behavioral: Personalized Technology Detailing
- Stigma Reduction + SBCM (Experimental)
  Interventions: Behavioral: HIV Stigma Reduction; Behavioral: Strengths-Based Case Management (SBCM)
- Stigma Reduction + Technology Detailing (Experimental)
  Interventions: Behavioral: HIV Stigma Reduction; Behavioral: Personalized Technology Detailing
- Stigma Reduction (Experimental)
  Interventions: Behavioral: HIV Stigma Reduction
- SBCM + Technology Detailing (Experimental)
  Interventions: Behavioral: Strengths-Based Case Management (SBCM); Behavioral: Personalized Technology Detailing
- SBCM (Experimental)
  Interventions: Behavioral: Strengths-Based Case Management (SBCM)
- Technology Detailing (Experimental)
  Interventions: Behavioral: Personalized Technology Detailing
- HIV Information Only (No Intervention): This arm will not receive any of the 4 intervention components but will receive information on successfully aging with HIV.

INTERVENTIONS:
Behavioral: Group-Based Social Support — This intervention involves weekly support group calls facilitated by a licensed counselor or therapist for 8 consecutive weeks. The calls will last approximately 90 minutes and will include 5-8 individuals per group. Groups will follow pre-determined topic areas, with participants encouraged to explore their feelings about the difficulties associated with normal aging, being HIV-positive, and living with HIV/AIDS as an older adult. Therapists will facilitate mutual support among group members, encourage greater openness and emotional expressiveness, and help participants to improve their social and family support and enhance their quality of life. This intervention is an adaptation of Telephone Supportive-Expressive Group Therapy (Heckman et al., 2013).
  Arms: Social Support; Social Support + SBCM; Social Support + SBCM + Technology Detailing; Social Support + Stigma Reduction; Social Support + Stigma Reduction + SBCM; Social Support + Stigma Reduction + SBCM + Tech Detailing; Social Support + Stigma Reduction + Technology Detailing; Social Support + Technology Detailing
Behavioral: HIV Stigma Reduction — This intervention involves weekly support group calls facilitated by a licensed counselor or therapist for 6 consecutive weeks. The calls will last approximately 60-90 minutes and will include 5-8 individuals per group. This intervention is grounded in minority stress theory and will use cognitive-behavioral strategies to help empower participants to cope with stressful and stigmatizing experiences. Intervention components may include minimizing self-stigmatizing attitudes, reducing engulfment, developing a sense of future and hope, and developing and pursuing meaningful life goals. This intervention is an adaptation of "Ending Self Stigma" (Lucksted et al., 2011).
  Arms: Social Support + Stigma Reduction; Social Support + Stigma Reduction + SBCM; Social Support + Stigma Reduction + SBCM + Tech Detailing; Social Support + Stigma Reduction + Technology Detailing; Stigma Reduction; Stigma Reduction + SBCM; Stigma Reduction + SBCM + Technology Detailing; Stigma Reduction + Technology Detailing
Behavioral: Strengths-Based Case Management (SBCM) — The investigators have adapted an individually-tailored strengths-based case management (SBCM) intervention to help address the multiple structural barriers faced by rural older PLH. The adapted intervention, delivered by trained research staff, will include two 60-minute telephone-based SBCM counseling sessions with shorter follow-up phone calls to check-in on progress and help patients navigate identified barriers. The case manager will provide tailored sessions based on individually-identified needs and proximal life stressors. Capitalizing on participants' personal strengths, case managers will help empower participants to navigate issues related to employment, insurance, mental health, housing, or transportation. This may include assistance understanding, applying for, and accessing benefits or programs.
  Arms: SBCM; SBCM + Technology Detailing; Social Support + SBCM; Social Support + SBCM + Technology Detailing; Social Support + Stigma Reduction + SBCM; Social Support + Stigma Reduction + SBCM + Tech Detailing; Stigma Reduction + SBCM; Stigma Reduction + SBCM + Technology Detailing
Behavioral: Personalized Technology Detailing — Participants will be called by a technology-fluent study staff member, who will assess the current state of their technology literacy, access, and use. Detailing will focus on advancing the participant along the technology use cascade (using the internet, possessing a device and service to access internet at home, using the internet to access their electronic health record and pharmacy services, seeking HIV-related information, and finding social support). Each participant will be provided with personalized assistance based on their local and personal circumstances. Because of the individualized advice provided, there will be a range of contacts between 1 and 5, at customized intervals. Detailing protocols include the option of providing the participant with a tablet including cellular service (for 3 months) when in-home internet service is not available or is cost prohibitive.
  Arms: SBCM + Technology Detailing; Social Support + SBCM + Technology Detailing; Social Support + Stigma Reduction + SBCM + Tech Detailing; Social Support + Stigma Reduction + Technology Detailing; Social Support + Technology Detailing; Stigma Reduction + SBCM + Technology Detailing; Stigma Reduction + Technology Detailing; Technology Detailing

SUMMARY:
Engagement in HIV medical care and adherence to HIV medications are both essential in improving health outcomes among people living with HIV (PLH), but PLH living in rural areas-who suffer higher mortality rates than their urban counterparts-can confront multiple barriers to care engagement and adherence, especially as they face the logistical, medical, and social challenges associated with aging. This project will pilot test four intervention components designed to improve care engagement and medication adherence to determine their impact on health outcomes and quality of life among rural, older PLH. The four intervention components, adapted from evidence-based interventions and delivered remotely, are: (1) counselor-facilitated peer social support, (2) HIV stigma reduction, (3) strengths-based case management, and (4) individually-tailored technology use optimization. The investigators hypothesize that components will be acceptable to participants, will be feasible to administer remotely, and will show preliminary impact on (1) the proportion of participants that have viral suppression and (2) health-related quality of life. Results from this study will provide us with tools to improve health outcomes for rural older people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or greater
* Living in a zip code classified as a "Small and Isolated Small Rural Town" area by Rural-Urban Commuting Area Codes (RUCAs), and/or in a county classified as rural based on RUCAs, and/or in a county with a score of .4 or higher on the index of relative rurality (IRR)
* Living in Alabama, Arkansas, Georgia, Kentucky, Mississippi, Missouri, Oklahoma, South Carolina, or Tennessee
* Living with HIV
* Indicates willingness to participate in support groups
* Indicates willingness to self-collect a dried blood spot sample
* Has a telephone at home
* Able to provide informed consent

Exclusion Criteria:

* Not meeting eligibility criteria described above

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, PhD, Principal Investigator — Center for AIDS Intervention Research, Medical College of Wisconsin; Andrew Petroll, MD, Principal Investigator — Center for AIDS Intervention Research, Medical College of Wisconsin
Locations (1):
- Center for AIDS Intervention Research, Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] O'Connell KA, Skevington SM. An international quality of life instrument to assess wellbeing in adults who are HIV-positive: a short form of the WHOQOL-HIV (31 items). AIDS Behav. 2012 Feb;16(2):452-60. doi: 10.1007/s10461-010-9863-0. PMID 21181253

RESULTS

PARTICIPANT FLOW:
Groups:
- Social Support + Stigma Reduction + SBCM + Tech Detailing: Group-Based Social Support Intervention + Group-Based HIV Stigma Reduction Intervention + Individual Strengths-Based Case Management Intervention + Individual Personalized Technology Detailing Intervention
- Social Support + Stigma Reduction + SBCM: Group-Based Social Support Intervention + Group-Based HIV Stigma Reduction Intervention + Individual Strengths-Based Case Management Intervention
- Social Support + Stigma Reduction + Technology Detailing: Group-Based Social Support Intervention + Group-Based HIV Stigma Reduction Intervention + Individual Personalized Technology Detailing Intervention
- Social Support + Stigma Reduction: Group-Based Social Support Intervention + Group-Based HIV Stigma Reduction Intervention
- Social Support + SBCM + Technology Detailing: Group-Based Social Support Intervention + Individual Strengths-Based Case Management Intervention + Individual Personalized Technology Detailing Intervention
- Social Support + SBCM: Group-Based Social Support Intervention + Individual Strengths-Based Case Management Intervention
- Social Support + Technology Detailing: Group-Based Social Support Intervention + Individual Personalized Technology Detailing Intervention
- Social Support: Group-Based Social Support Intervention
- Stigma Reduction + SBCM + Technology Detailing: Group-Based HIV Stigma Reduction Intervention + Individual Strengths-Based Case Management Intervention + Individual Personalized Technology Detailing Intervention
- Stigma Reduction + SBCM: Group-Based HIV Stigma Reduction Intervention + Individual Strengths-Based Case Management Intervention
- Stigma Reduction + Technology Detailing: Group-Based HIV Stigma Reduction Intervention + Individual Personalized Technology Detailing Intervention
- Stigma Reduction: Group-Based HIV Stigma Reduction Intervention
- SBCM + Technology Detailing: Individual Strengths-Based Case Management Intervention + Individual Personalized Technology Detailing Intervention
- SBCM: Individual Strengths-Based Case Management Intervention
- Technology Detailing: Individual Personalized Technology Detailing Intervention
Period: Overall Study
Arm/Group | Social Support + Stigma Reduction + SBCM + Tech Detailing | Social Support + Stigma Reduction + SBCM | Social Support + Stigma Reduction + Technology Detailing | Social Support + Stigma Reduction | Social Support + SBCM + Technology Detailing | Social Support + SBCM | Social Support + Technology Detailing | Social Support | Stigma Reduction + SBCM + Technology Detailing | Stigma Reduction + SBCM | Stigma Reduction + Technology Detailing | Stigma Reduction | SBCM + Technology Detailing | SBCM | Technology Detailing | HIV Information Only
Started | 4 | 4 | 3 | 3 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 2 | 4 | 2 | 3 | 2 | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Support + Stigma Reduction + SBCM + Tech Detailing | Social Support + Stigma Reduction + SBCM | Social Support + Stigma Reduction + Technology Detailing | Social Support + Stigma Reduction | Social Support + SBCM + Technology Detailing | Social Support + SBCM | Social Support + Technology Detailing | Social Support | Stigma Reduction + SBCM + Technology Detailing | Stigma Reduction + SBCM | Stigma Reduction + Technology Detailing | Stigma Reduction | SBCM + Technology Detailing | SBCM | Technology Detailing | HIV Information Only | Total
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [51 to 55.25] | 59 [56.75 to 61.25] | 55 [53 to 58] | 52 [51.5 to 52.5] | 54.5 [51.75 to 59.25] | 54 [53 to 57] | 59.5 [57 to 62.75] | 61 [50 to 72] | 55 [50.75 to 59.25] | 62 [56.5 to 66.5] | 61 [59.5 to 63.5] | 62 [60.25 to 64.25] | 61 [59.25 to 63.5] | 58.5 [56.5 to 60] | 54 [51.75 to 58.5] | 55 [53.5 to 56.75] | 57 [52 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 15
  Male | 2 | 4 | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2 | 3 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, Non-Hispanic | 1 | 3 | 2 | 2 | 2 | 4 | 4 | 1 | 1 | 2 | 3 | 2 | 4 | 2 | 2 | 4 | 39
  Race/Ethnicity: Black or African American or Caribbean, Non-Hispanic | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 19
  Race/Ethnicity: Latino/Hispanic, Any Race | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With HIV Viral Load ≥832 Copies/mL (HemaSpot DBS)
Description: Proportion of participants with HIV viral load ≥832 copies/mL, as measured through use of HemaSpot dried blood spot (DBS) testing. At baseline and follow-up, participants were sent dried blood spot (DBS) kits by mail to complete self-collection of blood samples for HIV viral load testing. Following specimen collection, participants placed the filled HemaSpot container into the shipping envelope, which sent the specimen directly to the clinical laboratory for testing. HemaSpot devices with sufficient blood volume were tested using Abbott m2000 RealTime HIV-1 dried blood spot (DBS) quantitative assay, with 832 copies/mL limit of detection. DBS viral load results were classified in three categories: 1. Detected and quantifiable at ≥832 copies/mL; 2. Detected and non-quantifiable, estimated between <832 and >300 copies/mL; and 3. Not detected, estimated to be <300 copies/mL.
Time Frame: 3 months following enrollment/baseline survey
Population: Analysis included all participants with follow-up HemaSpot DBS data (N = 49). Participants were included in outcome analyses in assigned arm regardless of intervention participation/attendance.
Measure: Count of Participants; unit: Participants
Groups:
- Social Support Intervention: Yes: Those randomized to group-based social support intervention.
- Social Support Intervention: No: Those not randomized to group-based social support intervention.
- Stigma Reduction Intervention: Yes: Those randomized to group-based stigma reduction intervention.
- Stigma Reduction Intervention: No: Those not randomized to group-based stigma reduction intervention.
- Strengths-Based Case Management Intervention: Yes: Those randomized to individual strengths-based case management intervention.
- Strengths-Based Case Management Intervention: No: Those not randomized to individual strengths-based case management intervention.
- Technology Detailing Intervention: Yes: Those randomized to individual personalized technology detailing intervention.
- Technology Detailing Intervention: No: Those not randomized to individual personalized technology detailing intervention.
Arm/Group | Social Support Intervention: Yes | Social Support Intervention: No | Stigma Reduction Intervention: Yes | Stigma Reduction Intervention: No | Strengths-Based Case Management Intervention: Yes | Strengths-Based Case Management Intervention: No | Technology Detailing Intervention: Yes | Technology Detailing Intervention: No
Number analyzed (Participants) | 22 | 27 | 24 | 25 | 24 | 25 | 27 | 22
Participants | 5 | 7 | 8 | 4 | 6 | 6 | 8 | 4
Statistical Analysis 1: Comparison: Social Support Intervention: Yes vs Social Support Intervention: No; We fit a generalized linear mixed model using the glmer function and a logit link in the R package lme4. The model included a random effect for participant. Predictors (fixed effects) included time (baseline vs. follow-up), random assignments, and interactions between assignments and time. We adjusted for mode of survey completion. Significant interactions indicated differential changes in outcomes over time for those randomly assigned vs. not randomly assigned to different interventions; Test type: Superiority; p = .33, Mixed Models Analysis — All tests performed were 2-sided. Given that the study was a pilot, we used α = .25 as a significance level cutoff and focus primarily on patterns in the data and effect sizes; Odds Ratio (OR) = 3.23
Statistical Analysis 2: Comparison: Stigma Reduction Intervention: Yes vs Stigma Reduction Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .63, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.76
Statistical Analysis 3: Comparison: Strengths-Based Case Management Intervention: Yes vs Strengths-Based Case Management Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .78, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.68
Statistical Analysis 4: Comparison: Technology Detailing Intervention: Yes vs Technology Detailing Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .90, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.87
Statistical Analysis 5: Comparison: Social Support Intervention: Yes; Given that our factorial design resulted in many "control" participants who were assigned to alternative interventions, for this pilot we also report on changes over time in outcomes for participants randomly assigned to each intervention. These changes tested with mixed models that contained only participants assigned to each intervention. Here, time was the predictor of interest, and we again controlled for mode of survey administration; Test type: Other — Single group change over time; p = .38, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.89
Statistical Analysis 6: Comparison: Stigma Reduction Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .78, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.25
Statistical Analysis 7: Comparison: Strengths-Based Case Management Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.32
Statistical Analysis 8: Comparison: Technology Detailing Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .91, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.92

2. Primary Outcome: Health-Related Quality of Life
Description: Based on full scale scores from the 31-item WHOQOL-HIV BREF (O'Connell & Skevington, 2012), with scores ranging from 0 to 100. Higher scores indicate higher (better) quality of life.
  Quality of life was assessed with 31 items from the WHOQOL-HIV BREF (O'Connell & Skevington, 2012). Domains assessed include physical health; psychological health; level of independence; social relationships; environmental health; and personal beliefs. Additionally, two individual items focus on overall quality of life and general health. Domain scores were created as described by the WHO, and we created a composite quality of life score by equally weighting the 6 domains, overall quality of life item, and general health item. The composite score was rescaled such that overall scores ranged from 0 to 100, with higher scores indicating better health-related quality of life.
Time Frame: 3 months following enrollment/baseline survey
Population: Analysis included all participants with follow-up survey data (N = 51). Participants were included in outcome analyses in assigned arm regardless of intervention participation/attendance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Support Intervention: Yes | Social Support Intervention: No | Stigma Reduction Intervention: Yes | Stigma Reduction Intervention: No | Strengths-Based Case Management Intervention: Yes | Strengths-Based Case Management Intervention: No | Technology Detailing Intervention: Yes | Technology Detailing Intervention: No
Number analyzed (Participants) | 24 | 27 | 26 | 25 | 26 | 25 | 28 | 23
score on a scale | 68.54 (15.37) | 64.97 (15.32) | 65.83 (13.96) | 67.51 (16.82) | 66.50 (16.75) | 66.81 (13.96) | 68.01 (15.64) | 65.00 (15.04)
Statistical Analysis 1: Comparison: Social Support Intervention: Yes vs Social Support Intervention: No; We fit a linear mixed model using the lmer function in the R package lme4. The model included a random effect for participant and utilized all available data. Predictors (fixed effects) included time (baseline vs. follow-up), random assignments, and interactions between assignments and time. We adjusted for mode of survey completion. Significant interactions indicated differential changes in outcomes over time for those randomly assigned vs. not randomly assigned to different interventions; Test type: Superiority; p = .36, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 2.58, Standard Error of Mean 2.80
Statistical Analysis 2: Comparison: Stigma Reduction Intervention: Yes vs Stigma Reduction Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .88, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -0.42, Standard Error of Mean 2.78
Statistical Analysis 3: Comparison: Strengths-Based Case Management Intervention: Yes vs Strengths-Based Case Management Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .89, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 0.38, Standard Error of Mean 2.80
Statistical Analysis 4: Comparison: Technology Detailing Intervention: Yes vs Technology Detailing Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .73, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -0.99, Standard Error of Mean 2.78
Statistical Analysis 5: Comparison: Social Support Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 4.88, Standard Error of Mean 1.83
Statistical Analysis 6: Comparison: Stigma Reduction Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .12, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 3.28, Standard Error of Mean 2.03
Statistical Analysis 7: Comparison: Strengths-Based Case Management Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 3.82, Standard Error of Mean 2.06
Statistical Analysis 8: Comparison: Technology Detailing Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .12, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 3.19, Standard Error of Mean 1.99

3. Secondary Outcome: Medication Adherence
Description: Adherence to HIV antiretroviral medications in the past 30 days was assessed with the 3 items from the Wilson adherence scale (Wilson et al., 2017; αs = .71-.79). This scale was scored in line with Wilson et al., with scores ranging from 0 to 100 and higher scores indicating better adherence. Due to significant skew in this outcome, we created a binary variable indicating perfect adherence to HIV medications.
Time Frame: 3 months following enrollment/baseline survey
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Social Support Intervention: Yes | Social Support Intervention: No | Stigma Reduction Intervention: Yes | Stigma Reduction Intervention: No | Strengths-Based Case Management Intervention: Yes | Strengths-Based Case Management Intervention: No | Technology Detailing Intervention: Yes | Technology Detailing Intervention: No
Number analyzed (Participants) | 24 | 27 | 26 | 25 | 26 | 25 | 28 | 23
Participants | 13 | 14 | 13 | 14 | 14 | 13 | 14 | 13
Statistical Analysis 1: Comparison: Social Support Intervention: Yes vs Social Support Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .049, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 22.30
Statistical Analysis 2: Comparison: Stigma Reduction Intervention: Yes vs Stigma Reduction Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .66, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.86
Statistical Analysis 3: Comparison: Strengths-Based Case Management Intervention: Yes vs Strengths-Based Case Management Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .78, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.68
Statistical Analysis 4: Comparison: Technology Detailing Intervention: Yes vs Technology Detailing Intervention: No; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.43
Statistical Analysis 5: Comparison: Social Support Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .09, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.26
Statistical Analysis 6: Comparison: Stigma Reduction Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .40, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.05
Statistical Analysis 7: Comparison: Strengths-Based Case Management Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .66, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.42
Statistical Analysis 8: Comparison: Technology Detailing Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .87, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.14

4. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms during the past 2 weeks were assessed with the 9 items from the Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001; αs = .87-.90). Participants indicated how often they had experienced different depressive symptoms (e.g., "Feeling down, depressed, or hopeless"). Responses ranged from not at all (0) to nearly every day (3). Items were summed to yield scores ranging from 0 to 27, with higher scores indicating more depressive symptoms.
Time Frame: 3 months following enrollment/baseline survey
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Support Intervention: Yes | Social Support Intervention: No | Stigma Reduction Intervention: Yes | Stigma Reduction Intervention: No | Strengths-Based Case Management Intervention: Yes | Strengths-Based Case Management Intervention: No | Technology Detailing Intervention: Yes | Technology Detailing Intervention: No
Number analyzed (Participants) | 24 | 27 | 26 | 25 | 26 | 25 | 28 | 23
score on a scale | 6.84 (6.62) | 9.33 (6.74) | 8.47 (6.59) | 7.84 (7.00) | 8.08 (7.32) | 8.25 (6.22) | 7.50 (7.43) | 8.96 (5.84)
Statistical Analysis 1: Comparison: Social Support Intervention: Yes vs Social Support Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .24, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -1.74, Standard Error of Mean 1.47
Statistical Analysis 2: Comparison: Stigma Reduction Intervention: Yes vs Stigma Reduction Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .17, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -2.05, Standard Error of Mean 1.46
Statistical Analysis 3: Comparison: Strengths-Based Case Management Intervention: Yes vs Strengths-Based Case Management Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .66, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = 0.64, Standard Error of Mean 1.47
Statistical Analysis 4: Comparison: Technology Detailing Intervention: Yes vs Technology Detailing Intervention: No; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .89, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -0.21, Standard Error of Mean 1.46
Statistical Analysis 5: Comparison: Social Support Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -1.60, Standard Error of Mean 0.75
Statistical Analysis 6: Comparison: Stigma Reduction Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .07, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -1.81, Standard Error of Mean 0.95
Statistical Analysis 7: Comparison: Strengths-Based Case Management Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .57, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -0.51, Standard Error of Mean 0.88
Statistical Analysis 8: Comparison: Technology Detailing Intervention: Yes; [analysis description as in outcome 1, analysis 5]; Test type: Other — Single group change over time; p = .42, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; B = -0.92, Standard Error of Mean 1.12

ADVERSE EVENTS:
Time Frame: Entire study period (an average of 126 days)
Arm/Group | Social Support + Stigma Reduction + SBCM + Tech Detailing | Social Support + Stigma Reduction + SBCM | Social Support + Stigma Reduction + Technology Detailing | Social Support + Stigma Reduction | Social Support + SBCM + Technology Detailing | Social Support + SBCM | Social Support + Technology Detailing | Social Support | Stigma Reduction + SBCM + Technology Detailing | Stigma Reduction + SBCM | Stigma Reduction + Technology Detailing | Stigma Reduction | SBCM + Technology Detailing | SBCM | Technology Detailing | HIV Information Only
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT04549259/Prot_SAP_000.pdf